CLINICAL TRIAL: NCT06853418
Title: Paired Non-inferiority Study Comparing Overture Semi-automated Vitrification System ("DaVitri") to Standard Manual Process for Clinical Pregnancy Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Overture Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP-DV-000-GEN-004
Record Dates: First submitted 2024-09-07; First posted 2025-03-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Oocyte Cryopreservation
Keywords: vitrification; oocytes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Manually vitrified oocytes (No Intervention): Control oocytes will be manually vitrified and placed into cryogenic storage.
- Test Oocytes (Experimental): Test oocytes will be prepared for vitrification using the DaVitri system. Following preparation with DaVitri, test oocytes will be loaded onto a cryogenic device that is placed into cryogenic storage.
  Interventions: Device: Oocyte Cryopreservation

INTERVENTIONS:
Device: Oocyte Cryopreservation — The DaVitri System is intended to semi-automate vitrification preparation of human oocytes.
  The Overture Semi-Automated Vitrification System ("DaVitri") is a medical device that uses semi-automated oocyte vitrification.
  The system comprises the DaVitri Station, and the DaVitri Dish. The DaVitri Station is a piece of capital equipment with touch screen control that manages the vitrification preparation. The DaVitri Dish is a cartridge-like device onto which oocytes and vitrification reagents are loaded. When the DaVitri Dish is loaded into the DaVitri Station, and the cryo process is initiated, a microfluidic pump controls the flow of reagents to and from the DaVitri Dish containing the oocytes.
  Arms: Test Oocytes

SUMMARY:
This study will recruit 260 female recipients (and up to a maximum of 130 donors). This study is a sequel to the protocol CP-DV-000-GEN-003, entitled, "NON-INFERIORITY STUDY COMPARING OVERTURE SEMI-AUTOMATED VITRIFICATION SYSTEM ("DaVitri") TO STANDARD MANUAL PROCESS USING BLASTOCYST RATE AS THE PRIMARY END POINT".

Donors will provide informed consent and will be enrolled before egg retrieval. Once the oocytes are retrieved, they will undergo thorough denudation to remove corona cells and will be assessed for maturity. Subsequently, mature MII oocytes exhibiting good morphology, as per the Vienna Consensus, ranging between 12 and 30 in number, will be processed.

These oocytes will then be randomly divided into groups comprising 6 to 8 oocytes each. Therefore, from a single donor, 2 to 4 groups can be generated. An identifier will be assigned for each group. One of the groups will be randomly selected. This group will be randomly assigned to DaVitri or Control. The remaining groups will be randomly selected and assigned alternatively to Control and DaVitri groups:

Control oocytes will be manually vitrified and placed into cryogenic storage. Test oocytes will be prepared for vitrification using the DaVitri system. Following preparation with DaVitri, test oocytes will be loaded onto a cryogenic device that is placed into cryogenic storage.

The same preservation media (Kitazato) will be used to prepare all oocytes.

All oocytes will be warmed manually. Survival rate will be recorded following warming. After warming, the oocytes will be fertilized via Intracytoplasmic Sperm Injection (ICSI) with either donor or patient's partner sperm and resulting embryos cultured to blastocyst stage, keeping score of which embryos come from the Test or Control group. Fertilization rate will be recorded.

Embryos will be morphologically assessed (according to Gardner grading system) on day 5-6 to determine blastulation rates and embryo quality in both groups. All the embryos will be vitrified according to the clinic's routine process and stored for further recipients.

Recipients will provide informed consent and will be enrolled before the retrieval of donor eggs. Once the donor has been matched with the recipient according to the phenotypic, demographic characteristics (following the regular clinical process established in the clinic donation program), the group of oocytes assigned will be randomly selected from either the DaVitri processed group or the manually processed group. Recipients of donated eggs will receive a single embryo transfer (SET).

The primary endpoint is Clinical Pregnancy Rate. Clinical Pregnancy will be confirmed by the presence of sac in uterus and chemical confirmation at 6-7 weeks after embryo transference, via ultrasound. Only the first embryo transfers will be used to calculate the primary endpoint. Successive transfers of any embryo group will not be considered inside the study.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria (donors) Ages 18-35 AMH range (2-10) ng/ml Healthy females (no pre-existing medical conditions)

Inclusion Criteria (recipient) Undergoing an in-vitro fertilization (IVF) cycle with egg donation Premenopausal female, 18-45 years of age Normal uterine cavity Single embryo transfer

Exclusion Criteria:

- Exclusion Criteria (donors) Age >35 years of age BMI <18.5 or >25 Infertility history Three previously failed IVF cycles, including abortions. Abnormal ovulation cycle FSH >10 or AMH <2 Alcoholism, drug addiction Infectious diseases (such as HIV, hepatitis, sexually transmitted infections) Donors producing less than 12 mature oocytes of good quality (according to Vienna Consensus criteria)

Sperm Exclusion Criteria Severe male factor Infertility (unless donated sperm is used) Alcoholism, drug addiction

Exclusion Criteria (recipients) Age >45 years of age BMI <18.5 or >29 Patients using a surrogate. Evidence of uterine pathologies Severe male factor Infertility (unless donated sperm is used) Alcoholism, drug addiction Infectious diseases (such as HIV, hepatitis, sexually transmitted infections)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | From enrollment to 6-7 weeks
  Presence of sac in uterus and chemical confirmation at 6-7 weeks

SECONDARY OUTCOMES:
Warming survival rates of oocytes | From enrollment to 2 weeks
  Vitrified and warmed Oocytes in this study will be evaluated for survival rates post warming. A skilled embryologist will evaluate survival based on a morphological assessment performed under a microscope. Warmed oocytes are considered to have survived if oocytes demonstrate the following characteristics:
  Expansion of oocyte, No dark/degenerated or contracted ooplasm No cracked zona pellucida
Fertilization Rates | From enrollment to 2 weeks
  Oocytes collected will be fertilized via Intracytoplasmic Sperm Injection (ICSI) where a single sperm cell is directly injected into the oocyte. Fertilization will be confirmed via the observation of two polar nuclear bodies (2PN) 18h
Gardner Score | From enrollment to 2 weeks
  This score will assess embryo quality based on the trophectoderm (TE) and inner cell mass (ICM). The resulting assessment will categorize embryos into two groups: non-viable embryos with very low implantation potential (DX, XD and DD embryo
Blastocyst Formation | From enrollment to 2 weeks
  Rates Fertilized oocytes (as confirmed via 2PN) will be cultured in an incubator for 5-7 days up to blastocyst stage. The number of fertilized oocytes which survive to the blastocyst stage will determine the blastocyst formation rate
Implantation rate | From enrollment to 3 weeks
  Embryos selected for transfer will be monitored for implantation. Implantation rate will be determined via a serum pregnancy test for human chorionic gonadotropin (hCG) 9-11 days post transference.
On-going pregnancy rate | From enrollment to 12 weeks
  12 weeks post transference the pregnancy rate will be evaluated by the presence of fetal heartbeat. It will confirm the absence of abortions. This heartbeat will be evaluated by ultrasound echography.
Congenital abnormality rate | From enrollment to 9 months
  Congenital abnormalities, also known as birth defects, are structural or functional abnormalities present at birth that can affect various parts of the body. The congenital abnormality rate will be measured for each group and
Delivery success rate | From enrollment to 9 months
  This rate is calculated by dividing the number of successful deliveries (live births) by the total number of treatment cycles or procedures performed, and then multiplying by 100 to express it as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Lane Fertility Institute, Novato, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.